CLINICAL TRIAL: NCT03623438
Title: Self-administered Acupressure for Insomnia Disorder: A Randomized Controlled Trial
Brief Title: Self-administered Acupressure for Insomnia Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SelfAcupInsomnia
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2019-10

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-administered acupressure group (Experimental): Subjects will attend two weekly 120-minute of self-administered acupressure training
  Interventions: Behavioral: Self-administered acupressure group
- Sleep hygiene education (SHE) group (Active Comparator): Subjects will attend two weekly 120-minute of sleep hygiene education
  Interventions: Behavioral: Sleep hygiene education (SHE) group

INTERVENTIONS:
Behavioral: Self-administered acupressure group — Subjects in the self-administered acupressure group will attend an acupressure training course (2 sessions, 2 hours each) to learn self-administered acupressure, which will then be performed every night for 4 weeks.
  Arms: Self-administered acupressure group
Behavioral: Sleep hygiene education (SHE) group — Subjects in the comparison group will receive sleep hygiene education (2 sessions, 2 hours each, same as the treatment group) and be reminded to follow the sleep hygiene practice daily for 4 weeks.
  Arms: Sleep hygiene education (SHE) group

SUMMARY:
The study is to evaluate the clinical effects of self-administered acupressure for treating insomnia disorder delivered by a training course. Subjects will be offered either self-administered acupressure training or sleep hygiene education. Their insomnia severity will be compared after 8 weeks.

DETAILED DESCRIPTION:
Objectives: To evaluate the clinical effects of self-administered acupressure for treating insomnia disorder delivered by a training course.

Hypothesis: Subjects in the self-administered acupressure group will have greater improvement in insomnia symptoms and daytime impairment than those in the sleep hygiene education (SHE) group at 4 weeks and 8 weeks.

Design and subjects: A randomized controlled trial. 184 subjects with insomnia disorder recruited from the community will be randomized to self-administered acupressure or SHE groups in a 1: 1 ratio.

Study instrument: Insomnia Severity Index (ISI) will be used to assess insomnia symptoms and daytime impairment.

Interventions: Subjects in the self-administered acupressure group will attend two training lessons (2-hour each) to learn self-administered acupressure and practice it every night for 4 weeks; subjects in the SHE group will receive sleep hygiene education with the schedule and duration that are same to the self-administered acupressure group.

Main outcome measures: The primary outcome measure is the ISI score. Other measures include sleep parameters by subjective sleep diary and objective actigraphy, Hospital Anxiety and Depression Scale, and SF-6D at 4 and 8 weeks. Acceptability and compliance of self-administered acupressure will be evaluated.

Data Analysis: Differences in the questionnaire scores, subjective and objective sleep parameters will be examined using a mixed-effects model.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese Hong Kong residents who are able to communicate in Cantonese or Putonghua;
2. Aged 18-64 years;
3. A current clinical DSM-5 diagnosis of insomnia disorder according to the Brief Insomnia Questionnaire (BIQ)
4. Insomnia Severity Index total score of at least 10 indicating insomnia at the clinical level; and
5. Willing to give informed consent and comply with the trial protocol.

Exclusion Criteria:

1. Receiving acupuncture or practitioner-delivered acupressure treatment in the past 6 months;
2. Pregnancy;
3. Cognitive impairment as indicated by a Mini Mental State Examination ≤23;
4. At significant suicidal risk as rated by the Hamilton Depression Rating Scale item on suicide (score ≥3) ;
5. No comorbid sleep disorders primarily requiring other treatment, such as sleep apnea or narcolepsy;
6. Taking herbal remedies, over-the-counter medication, or psychotropic drugs that target insomnia within the 2 weeks prior to baseline; and
7. Shift-workers/

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Week 8
  The ISI is a seven-item self-rating scale. The subjects rate the severity of insomnia, distress and functional impairment associated with insomnia on a 5-point Likert scale. The total score will be reported. The score ranges from 0 to 28; a higher score indicates a more severe condition.

SECONDARY OUTCOMES:
The 7-day daily sleep diary | Baseline, Week 4, Week8
  The standardized sleep diary records the daily sleep parameters.
Hospital Anxiety and Depression Scale (HADS) | Baseline, Week 4, Week8
  The HADS is a 14-item self-administrated questionnaire, which assesses the severity of depressive and anxiety symptoms. The anxiety and depression subscore will be reported. The subscore ranges from 0 to 21; a higher score indicates a more severe condition.
The 7-day actigraphy | Baseline, Week 4, Week8
  An actigraph is a watch-like device used to estimate sleep-wake schedules by measuring activity.
Short Form- 6 Dimensions | Baseline, Week 4, Week8
  It is a preference-based measure of health derived from the Short Form-36. It includes six dimensions: physical functioning, role participation, social functioning, bodily pain, mental health, and vitality. The total score will be reported. The score ranges from 0 to 1; a higher score indicates a better outcome.

OTHER OUTCOMES:
Credibility of Treatment Rating Scale | Baseline
  The 4-item Credibility of Treatment Rating Scale will be used to assess subjects' expectation towards the intervention in both groups. The score of each item will be reported. The score of each item ranges from 1 to 6. A higher score indicates a higher confidence toward the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, the Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Upon request